CLINICAL TRIAL: NCT02165033
Title: Multiple-dose Pharmacokinetics and Tolerability of "SYN006 HFA MDI" (Budesonide 180ug + Procaterol Hydrochloride 10ug/Dose HFA MDI) Administered Orally to Healthy Volunteers
Brief Title: Multiple-dose Pharmacokinetics Study of "SYN006 HFA MDI" Administered Orally to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCPK10002J1
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Budesonide/Procaterol 180/10 X 4 puffs (Experimental): Multiple dose of SYN006 HFA MDI (Budesonide 180ug + Procaterol 10ug/puff), 4 puffs each day for consecutive 7 days
  Interventions: Drug: Budesonide/Procaterol 180/10 X 4 puffs

INTERVENTIONS:
Drug: Budesonide/Procaterol 180/10 X 4 puffs — Budesonide/Procaterol 180/10mcg, 4 puffs, Repeated dose
  Other Names: SYN006 HFA MDI

SUMMARY:
Budesonide + Procaterol HFA MDI is a novel asthma product containing both budesonide and procaterol in a single inhaler. Budesonide is a corticosteroid that treats underlying airway inflammation in asthma. Procaterol is a direct acting sympathomimetic with predominantly Beta-adrenoceptor stimulant activity selective to Beta-2 receptors (a Beta-2 agonist). It is used as a bronchodilator in the management of reversible airways obstructive pulmonary disease. Budesonide and Procaterol therefore have complementary effects, treating two different components of asthma.

DETAILED DESCRIPTION:
Test drug: SYN006 HFA MDI Batch No: BPP-033-088 Dosage Form: HFA Metered Dose Inhaler Active Substance: Budesonide 180ug and procaterol hydrochloride hydrate 10ug/dose Dosage regimen: Multiple dose (4 puffs: budesonide 720ug and procaterol hydrochloride hydrate 40ug); thirteen consecutive doses

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
* Healthy adults, aged between 20 and 40 years old.
* Subjects with Body Mass Index (BMI) of >=18.5 and <=25.0 (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2]).
* Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest x-ray and electrocardiogram.
* Clinical laboratory test: within limit of normal range or acceptable to investigator.

Exclusion Criteria:

* History of drug or alcohol abuse within the past year.
* Medical history of severe drug allergy or sensitivity to analogous drug.
* Evidence of acute or chronic diseases or having undergone surgery from 4 weeks prior to Period I dosing.
* Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology. Creatinine > 2UNL (upper normal limit); Liver enzymes > 2UNL; Total bilirubin > 2UNL.
* Planned vaccination during the time course of the study.
* Taking any clinical investigation drug from 2 months prior to Period I dosing.
* Use of any medication, including herb medicine from 4 weeks before dosing.
* Donation of 500mL of blood in the past 3 months prior to dosing or donation of 250mL of blood in the past 2 months prior to dosing.
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result.
* A positive test for HIV antibody.
* In screening subjects will be given training to ensure that subjects are able to correctly use the investigational products. If the subjects, the use of the investigational products lack of proficiency will not be included in this study.
* Students of National Defense Medical Center.
* For female subjects, if they meet any of the following criteria:

  1. Lactating women
  2. Positive pregnancy test (urine) at screening, or prior to dosing
  3. Do not use adequate contraception during the study
  4. Women taking oral contraceptives

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) at day 1 | predose,0.083,0.167,0.333,0.5,0.75,1,1.5,2,3,4,6,8,10,12 hours post-dose
Peak Plasma Concentration (Cmax) at day 1 | predose,0.083,0.167,0.333,0.5,0.75,1,1.5,2,3,4,6,8,10,12 hours post-dose
Tmax at day 1 | predose,0.083,0.167,0.333,0.5,0.75,1,1.5,2,3,4,6,8,10,12 hours post-dose
Area Under Curve (AUC) at day 7 | predose,0.083,0.167,0.333,0.5,0.75,1,1.5,2,3,4,6,8,10,12 hours post-dose
Peak Plasma Concentration (Cmax) at day 7 | predose,0.083,0.167,0.333,0.5,0.75,1,1.5,2,3,4,6,8,10,12 hours post-dose
Tmax at day 7 | predose,0.083,0.167,0.333,0.5,0.75,1,1.5,2,3,4,6,8,10,12 hours post-dose

SECONDARY OUTCOMES:
Accumulation ratio of AUC at day 1 and day 7 | 0.083, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: C W Perng, M.D, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan